CLINICAL TRIAL: NCT06154993
Title: Comparison of Static and Dynamic Opening With Neural Sliding in Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S22C08G30001
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cervical; Cervical Radiculopathy
Keywords: cervical radiculopathy; static opener; dynamic opener; slider neurodynamic
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- static opener with slider + Conventional PT (Experimental): Patient supine Maintaining neck flexion + contralateral flexion and rotation and applying median nerve slider mobilization while maintaining the neck static in mentioned position.
  Conventional PT includes hot pack for 10 mins and cervical isometrics.
  Interventions: Other: static opening with slider+ Conventional PT
- dynamic opener with slider + Conventional PT (Experimental): Patient supine Neck flexion + contralateral flexion and rotation. And sliding the median nerve along with neck movement from contralateral flexion+rotation to neutal position in repetitive manner, by releasing tension from median nerve when bringing neck in neutral to ease tension from affected side.
  Conventional PT includes hot pack for 10 mins and cervical isometrics.
  Interventions: Other: dynamic opener with slider + Conventional PT

INTERVENTIONS:
Other: static opening with slider+ Conventional PT — Patient supine Maintaining neck flexion + contralateral flexion and rotation and applying median nerve slider mobilization while maintaining the neck static in mentioned position.
  Frequency: 3 sets of 10 reps with 5 sec hold for 3 times/week for 4 weeks Conventional PT includes hot pack for 10 mins and cervical isometrics. Frequency: 3 sets of 10 reps with 5 sec hold for 3 times/week for 4 weeks.
  Duration: 30-40 mins
  Arms: static opener with slider + Conventional PT
Other: dynamic opener with slider + Conventional PT — Patient supine Neck flexion + contralateral flexion and rotation. And sliding the median nerve along with neck movement from contralateral flexion+rotation to neutal position in repetitive manner, by releasing tension from median nerve when bringing neck in neutral to ease tension from affected side.
  Conventional PT includes hot pack for 10 mins and cervical isometrics. Frequency: 3 sets of 10 reps with 5 sec hold for 3 times/week for 4 weeks.
  Duration: 30-40 mins
  Arms: dynamic opener with slider + Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to determine the effects of static and dynamic opening with neural sliding in patients with cervical radiculopathy for reducing pain, enhancing cervical range of motion and improve functional status.

DETAILED DESCRIPTION:
Static opener is a neurodynamic technique for cervical radiculopathy for reducing pressure on the nervous system that causes intervertebral foramina to remain in the open position for a certain period. This enables blood flow to return to neural tissue so that oxygenation is improved, along with slider mobilization will reduce symptoms and give better healing to the inflamed nerve. when the intervertebral foramina remain open for a considerable amount of time axoplasmic flow is reestablished, oxygenation is improved, increases blood flow along with venous return and nerve gets more nutrients and all the inflammatory exudate is taken off resulting for early improvement.

Dynamic opener is a neurodynamic technique in opening direction to repetitively open and close the intervertebral foramina and produces oscillatory movements that cause pumping effect on the nerve and help to drain edema due to inflammation and help reduce pain and increase the range also.

ELIGIBILITY:
Inclusion Criteria:

* : • Spurling +ive

  * Distraction test +ive (alleviate symptoms)
  * Pain, paresthesia and numbness in Rt/Lt UL in dermatomal pattern of median nerve
  * MRI confirmed spondylosis or disc herniation
  * Age 35-60

Exclusion Criteria:

* • Cervical spine fracture

  * RA
  * Cervical myelopathy
  * Systemic neurological conditions
  * Osteoporosis

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
neck disability index | 4 weeks
  Most used questionnaire for disability in patient related to any musculoskeletal neck condition. It has 7 items for daily living, 2 for pain and 1 for concentration. Each item is rated from 0 to 5. Total score is presented in percentage. Higher score tells greater disability while 0 means no disability. Total score is 50.
visual analogue scale | 4 weeks
  VAS is a commonly used assessment tool for pain intensity ranging from 0 to 100mm on a horizontal scale while patient marks a vertical line to rank his/her pain.
  0-4mm no pain 5-44mm mild pain 45-74mm moderate pain 75-100mm severe pain
inclinometer | 4 weeks
  A device used to check range of motion based on gravity.

CONTACTS AND LOCATIONS:
Overall Officials: Affan Iqbal, Phd*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - RehabWrox, Islamabad, Federal
  - Pakistan Railway General Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No